CLINICAL TRIAL: NCT06684392
Title: Assessment of the Effect of an Inspiratory Muscle Training Regimen on Decannulation Time in Adult Hospitalized Subjects with Tracheostomy Secondary to Prolonged Mechanical Ventilation
Brief Title: Assessment of the Effect of an Inspiratory Muscle Training Regimen on Decannulation Time in Tracheostomized Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Dr. Franco Ravera Zunino (Other)
Collaborators: University of Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FONIS2024
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Tracheostomy Complication; Diaphragm Disease
Keywords: tracheostomy; inspiratory muscle training; diaphragm dysfunction; diaphragm ultrasound

STUDY DESIGN:
Intervention Model Description: Control Group (CG): The CG will follow the current protocol at HRLBO. This involves a weaning protocol from mechanical ventilation 24 hours after tracheostomy placement. Initial disconnection windows are 2 hours in the morning and 2 hours in the afternoon. If tolerated, the next day's windows extend to 4 hours each, and by the third day, to 6 hours. On the fourth day, a continuous 12-hour disconnection is attempted, progressing to 24 if successful. Additionally, subjects will train at 50% of their MIP in 5 sets of 6 breaths once weaned.
  Intervention Group (IG): The IG will follow the CG protocol plus inspiratory muscle training (IMT). If weaning or disconnection is not achieved, subjects will train for inspiratory strength alone. Once weaning or disconnection is successful, the new IMT protocol combining strength and endurance training will begin. If the patient shows clinical signs of respiratory failure, IMT will be paused for the day.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): The control group will follow the current protocol at HRLBO. This involves a weaning protocol from mechanical ventilation 24 hours after tracheostomy placement. Initial disconnection windows are 2 hours in the morning and 2 hours in the afternoon. If tolerated, the next day's windows are extended to 4 hours each. On the third day, the windows are extended to 6 hours each. On the fourth day, a continuous 12-hour disconnection is attempted, progressing to 24 hours if successful. Additionally, subjects will train at 50% of their maximum inspiratory pressure (MIP) in 5 sets of 6 breaths once weaned from mechanical ventilation. If tracheostomy tube occlusion (defined as temporary closure of airflow through the tracheostomy tube, using physiological ventilation) is achieved for 24 hours and the decannulation criteria are met, the tracheostomy tube will be removed.
- Experimental Group (Experimental): The intervention group will follow the current HRLBO protocol, with the addition of an Inspiratory Muscle Training (IMT) regimen. Subjects will train only inspiratory muscle strength if they do not achieve weaning or complete disconnection from mechanical ventilation. Once they achieve weaning or disconnection, the new IMT regimen, combining strength and endurance training, will begin. On days when MIP evaluation is scheduled according to the IMT protocol, training time will be replaced by evaluation to avoid excessive ventilatory workload, limiting training to once a day. If a patient exhibits two or more clinical criteria for respiratory failure, IMT will be suspended for that day. These criteria include: RR > 35 bpm; SpO2 < 88%; HR > 130 bpm; SBP > 180 mmHg or < 90 mmHg; Modified Borg score > 6, signs of agitation, sweating, or altered consciousness.
  Interventions: Other: Inspiratory muscle training

INTERVENTIONS:
Other: Inspiratory muscle training — Subjects will train only inspiratory muscle strength if they do not achieve VP or definitive disconnection of MV, and, when they already achieve these VP or definitive disconnection, the new EMI regimen that combines strength and resistance training will begin to be applied. Inspiratory muscle training guideline (EMI). On the day that, according to the EMI guideline, the Pimax evaluation corresponds, the training time will be replaced by the evaluation to avoid overloading the subjects with ventilatory work, training them only once a day.
  Arms: Experimental Group

SUMMARY:
The objective of this project is to evaluate the effect of applying an individualized inspiratory muscle training regimen, combining strength and endurance exercises over a two-week period, on improving maximum inspiratory pressure, diaphragm thickness fraction, and its impact on successful decannulation time in patients with tracheostomy secondary to prolonged mechanical ventilation at HRLBO. Two groups of adult tracheostomized patients will be assessed: an experimental group, who will follow an individualized inspiratory muscle training regimen for 14 days along with standard physiotherapy, and a control group, who will receive standard physiotherapy and guided weaning through scheduled disconnection windows from mechanical ventilation. Both groups will be compared in terms of decannulation time, ICU length of stay, hospital days, and quality of life survey scores. The results of this study will help optimize the management of tracheostomized patients locally and nationally, reducing economic costs for both the country and the patients, and improving their quality of life, contributing to some health objectives for the 2011-2020 decade.

DETAILED DESCRIPTION:
Mechanical ventilation is a life-support intervention crucial for saving lives in ICU patients. However, its prolonged use leads to deterioration in respiratory muscle strength and endurance, causing diaphragm dysfunction. This weakening is associated with prolonged mechanical ventilation and increased difficulty in weaning the patient from the ventilator, known as "difficult weaning." It has been reported that up to 20% of ICU patients require tracheostomy due to this issue. Tracheostomy is an invasive procedure that involves creating an ostomy in the trachea to establish an artificial airway, allowing for ventilation, facilitating weaning from mechanical ventilation, and improving secretion management. However, muscle dysfunction from disuse and lack of effective respiratory muscle training extends the tracheostomy duration, leading to hospital-acquired infections, swallowing disorders, and increased ICU and hospital days. Thus, respiratory muscle training is a key tool for enabling tracheostomy removal (decannulation) and improving respiratory system efficiency. Since no universally accepted training protocol exists, it is not a common practice in ICUs worldwide, including our country. This project proposes that applying an individualized inspiratory muscle training regimen combining strength and endurance exercises for two weeks could improve respiratory muscle performance, reducing decannulation time (days from tracheostomy placement to removal).

The objective of this project is to assess the effect of an individualized inspiratory muscle training regimen, combining strength and endurance exercises for two weeks, on improving maximum inspiratory pressure, diaphragm thickness fraction, and its impact on successful decannulation time in patients with tracheostomy secondary to prolonged mechanical ventilation at HRLBO. Two groups of adult tracheostomized patients will be evaluated: an experimental group undergoing individualized inspiratory muscle training for 14 days plus standard physiotherapy, and a control group receiving standard physiotherapy and weaning guided by scheduled mechanical ventilation disconnection windows. Both groups will be compared in terms of decannulation time, ICU length of stay, hospital days, and quality of life survey scores. The study results will optimize the management of tracheostomized patients locally and nationally, reducing economic costs for both the country and patients and improving their quality of life, thus aiding in meeting some health objectives for the 2011-2020 decade.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients aged ≥ 18 years
* Connected to mechanical ventilation
* Secondary tracheostomy due to prolonged mechanical ventilation
* Glasgow Coma Scale (GCS) > 11 points
* Level of cooperation score (S5Q) > 3 points

Exclusion Criteria:

* Limitation of therapeutic effort (LTE*)
* Pregnancy
* Transfer to another center before completing the training (2 weeks)
* Degenerative neuromuscular disease
* Refusal to participate in this study (declining to provide informed consent [IC]).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Maximal inspiratory pressure | 2 weeks
  Maximum inspiratory pressure will be measured with the PowerBreathe valve before and after the training protocol to determine changes in diaphragm strength

SECONDARY OUTCOMES:
Diaphragm thickness | 2 weeks
  Changes in diaphragm thickness will be assessed via ultrasound before and after the training protocol.
Diaphragm excursion | 2 weeks
  Changes in diaphragm excursion will be assessed via ultrasound before and after the training protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Regional Franco Ravera Zunino, Rancagua, Región del Libertador General Bernardo O’Higgins, Chile

IPD SHARING:
Plan to Share IPD: Undecided